CLINICAL TRIAL: NCT00913055
Title: An Open-Label Study to Evaluate the Pharmacokinetic and Pharmacodynamic Response of a Hydrated and Non-Hydrated 84mg Octreotide Implant in Patients With Acromegaly
Brief Title: Open Label Study of Octreotide Implant in Patients With Acromegaly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Mark Roessel, Endo Pharmaceuticals Solutions
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-07-000
Record Dates: First submitted 2009-05-26; First posted 2009-06-03 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Acromegaly
Keywords: S-LAR; Octreotide; Implant
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One hydrated 84mg Octreotide implant (Experimental): hydrated implant
  Interventions: Drug: octreotide acetate
- One non-hydrated 84mg Octreotide implant (Experimental)
  Interventions: Drug: octreotide acetate

INTERVENTIONS:
Drug: octreotide acetate — subcutaneous implant

SUMMARY:
To evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) response of a hydrated and non-hydrated 84 mg octreotide implant in patients with acromegaly in the first 6 weeks of treatment.

DETAILED DESCRIPTION:
An open-label, randomized, multi-center, parallel-group, Phase I/II study conducted in 30 male and female patients with acromegaly. Eligible patients received 1 implant, either hydrated or non-hydrated, within 7 days of their Screening Visit. The octreotide implant was inserted subcutaneously in the inner aspect of their non-dominant arm under local anesthesia. Blood samples for the determination of insulin-like growth factor 1 (IGF-1), growth hormone (GH), and octreotide serum concentrations were collected at predetermined timepoints within the first 6 weeks after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with acromegaly
* Must be at least 18 years old
* Confirmed diagnosis of a growth hormone -secreting tumor
* Must be either a full or partial responder to octreotide demonstrated by historical laboratory values

Exclusion Criteria:

* Women who are pregnant, lactating or of child-bearing potential who are not practicing a medically acceptable method of birth control
* Patients with liver disease
* Patients with symptomatic cholelithiasis
* Patients receiving radiotherapy for their pituitary tumor at any time before Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)